CLINICAL TRIAL: NCT01819311
Title: Attention Bias Modification Training for Child Anxiety CBT Nonresponders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MH097931
Record Dates: First submitted 2013-03-12; First posted 2013-03-27 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-09

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Attention Bias Modification (Experimental): Attention Bias Modification is a computer-based attention training program
  Interventions: Behavioral: Attention Bias Modification
- Placebo Attention Task (Placebo Comparator): The Placebo Attention Task uses the same computer-based format and stimuli as the Attention Bias Modification Task, but does not train attention toward or away from stimuli.
  Interventions: Behavioral: Placebo Attention Task

INTERVENTIONS:
Behavioral: Attention Bias Modification — At each of eight sessions, participants complete 160 computer administered trials wherein a pair of threatening stimuli and neutral stimuli is presented simultaneously and then followed immediately by a probe. The probe always replaces the neutral stimulus and never replaces the threatening stimulus. The intervention is based on the idea that attention can be shaped via repetitive computer based training methods, and training attention toward neutral stimuli will lead to a reduction in anxiety and its disorders.
  Arms: Attention Bias Modification
Behavioral: Placebo Attention Task — At each of eight sessions, participants complete 160 computer administered trials wherein a pair of threatening stimuli and neutral stimuli is presented simultaneously and then followed immediately by a probe. The probe replaces the neutral stimulus and the threatening stimulus with equal probability.
  Arms: Placebo Attention Task

SUMMARY:
This project will test Attention Bias Modification Training (ABMT) among children and adolescents who have completed a full protocol of cognitive behavior therapy (CBT) for anxiety and still meet criteria for a primary diagnosis of an anxiety disorder. The purpose of this project is to determine whether ABMT leads to reductions in anxiety and related impairment, relative to a placebo task condition.

DETAILED DESCRIPTION:
This application proposes a pilot test of Attention Bias Modification Training (ABMT) among children and adolescents who have completed a full protocol of cognitive behavior therapy (CBT) for anxiety and still meet criteria for a primary diagnosis of an anxiety disorder a full year after completion of CBT. There is currently not a single empirical study in the youth anxiety treatment literature that has systematically examined a treatment augment for youth who fail to respond to a full course of CBT. Empirical efforts to address this issue are important because youths who do not respond to CBT continue to suffer emotional distress and impairment associated with anxiety disorders, experience frustration and demoralization by perceived "failure," and likely pose a financial burden on the health care system.

ABMT is a novel translational treatment for anxiety based on experimental and neuroscience research findings on attention processes. Research demonstrates that ABMT leads to reductions in anxiety and its disorders. Based on recent theory and research demonstrating an attention bias toward threat predicts CBT nonresponse among anxious youth, researchers have postulated that ABMT may hold promise as an augment to CBT because of its specific focus on attention bias that targets both frontal-cortical and subcortical circuitry.

This study will recruit an estimated 70 children and adolescents who have completed a 12-14 week CBT trial for anxiety disorders and at the one year follow-up continue to meet criteria for a primary diagnosis of an anxiety disorders. These 70 children and adolescents (ages 8-16 years) will be randomly assigned to complete eight biweekly sessions of either ABMT or a placebo control (PC) task. Clinician ratings on youth anxiety severity will be collected and evaluated as the primary outcome. Youth self ratings on anxiety symptoms and parent ratings on youth anxiety symptoms will be collected and evaluated as secondary outcomes. All measures will be collected before condition assignment (pretreatment), at immediate posttreatment, and at an eight week follow up. The following specific aims will be addressed.

Aim 1: Test whether ABMT leads to significantly lower levels of anxiety at posttreatment as compared to a Placebo Control Task.

Aim 2: Examine whether ABMT leads to significantly lower levels of anxiety as compared to a Placebo Control Task at a follow up evaluation eight weeks posttreatment. This would suggest the maintenance of ABMT effects after eight weeks of no treatment.

Aim 3: Gain perspective on the viability of variables as potential mediators and moderator of ABMT so as to inform decisions about whether to pursue these variables in a future R01. The variables proposed as potential mediators are attention bias toward threat and threat-related interpretation bias. The variable proposed as a potential moderator is attention control.

Overall, this project will provide critically needed data on ABMT as a treatment augment for youth with anxiety disorders who do not respond CBT. With these data in hand, the field will be in a better position to determine whether and how ABMT may be used optimally among anxious youth who are likely to need more than CBT.

ELIGIBILITY:
Inclusion Criteria:

* 8-16 years old
* completed a 12-14 week cognitive behavioral therapy for anxiety
* a primary DSM-IV diagnosis of generalized anxiety disorder, social anxiety disorder, or separation anxiety disorder
* if other psychiatric disorders are present, they must be treated with medication and stable

Exclusion Criteria:

* meet diagnostic criteria for Organic Mental Disorders, Psychotic Disorders, Pervasive Developmental Disorders, or Mental Retardation
* a high likelihood of harming self or others
* not been living with a primary caregiver for at least 6 months who is legally able to give consent for the child's participation
* previously undisclosed abuse requiring investigation or ongoing supervision by the Department of Social Services;
* involved currently in another psychosocial/behavioral treatment
* a serious vision problem that is not corrected with prescription lenses
* a physical disability that interferes with the ability to click a mouse button rapidly and repeatedly

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Pettit, PhD, Principal Investigator — Florida International University; Wendy Silverman, PhD, Principal Investigator — Yale Child Study Centery
Locations (1):
- Florida International University Center for Children and Families, Miami, Florida, United States

REFERENCES:
- [Derived] Pettit JW, Bechor M, Rey Y, Vasey MW, Abend R, Pine DS, Bar-Haim Y, Jaccard J, Silverman WK. A Randomized Controlled Trial of Attention Bias Modification Treatment in Youth With Treatment-Resistant Anxiety Disorders. J Am Acad Child Adolesc Psychiatry. 2020 Jan;59(1):157-165. doi: 10.1016/j.jaac.2019.02.018. Epub 2019 Mar 13. PMID 30877049

RESULTS

PARTICIPANT FLOW:
Period: Treatment Phase (4 Weeks)
Arm/Group | Attention Bias Modification | Placebo Attention Task
Started | 33 | 31
Completed | 31 | 30
Not Completed | 2 | 1
Period: Follow-up Phase (8 Weeks)
Arm/Group | Attention Bias Modification | Placebo Attention Task
Started | 31 | 30
Completed | 24 | 23
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Bias Modification | Placebo Attention Task | Total
Number analyzed (Participants) | 33 | 31 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.18 (2.69) | 11.26 (2.16) | 11.8 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 12 | 30
  Male | 15 | 19 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 27 | 55
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 28 | 27 | 55
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 2 | 0 | 2
Pediatric Anxiety Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Pediatric Anxiety Rating Scale (PARS) assesses global anxiety severity across social anxiety disorder, separation anxiety disorder, and generalized anxiety disorder in youth ages 6-17 years. An independent evaluator rates anxiety symptoms on 7 dimensions (i.e., number of symptoms, severity of distress, severity of physical symptoms, frequency, avoidance, interference at home, and interference out of home). Each dimension is rated from 0 to 5. Total scores range from 0 to 35, with higher scores indicating greater anxiety severity.
  units on a scale | 14.55 (3.63) | 13.12 (3.90) | 13.96 (3.84)
Screen for Child Anxiety and Related Emotional Disorders - Parent Version [Mean (Standard Deviation); unit: units on a scale] — The Screen for Child Anxiety Related Emotional Disorders - Parent Version (SCARED-P) assesses anxiety symptom severity in youth ages 6-17 years. The parent rates youth anxiety symptoms on 41 items; each item is rated from 0 to 2. Total scores range from 0 to 82, with higher scores indicating greater anxiety severity.
  units on a scale | 27.74 (14.57) | 26.24 (12.46) | 26.76 (13.68)
Screen for Child Anxiety and Related Emotional Disorders - Child Version [Mean (Standard Deviation); unit: units on a scale] — The Screen for Child Anxiety Related Emotional Disorders - Child Version (SCARED-C) assesses anxiety symptom severity in youth ages 6-17 years. The child rates his or her anxiety symptoms on 41 items; each item is rated from 0 to 2. Total scores range from 0 to 82, with higher scores indicating greater anxiety severity.
  units on a scale | 23.03 (12.81) | 22.87 (15.65) | 22.99 (14.92)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Rating on the Pediatric Anxiety Rating Scale
Description: The Pediatric Anxiety Rating Scale (PARS) assesses global anxiety severity across social anxiety disorder, separation anxiety disorder, and generalized anxiety disorder in youth ages 6-17 years. An independent evaluator rates anxiety symptoms on 7 dimensions (i.e., number of symptoms, severity of distress, severity of physical symptoms, frequency, avoidance, interference at home, and interference out of home). Each dimension is rated from 0 to 5. Total scores range from 0 to 35, with higher scores indicating greater anxiety severity.
Time Frame: post-treatment (within one week of completing the final of 8 semi-weekly sessions of Attention Bias Modification)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Bias Modification | Placebo Attention Task
Number analyzed (Participants) | 31 | 30
units on a scale | 8.88 (5.64) | 8.12 (5.03)

2. Primary Outcome: Clinician Rating on the Pediatric Anxiety Rating Scale
Description: as for outcome 1
Time Frame: 8-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Bias Modification | Placebo Attention Task
Number analyzed (Participants) | 24 | 23
units on a scale | 9.50 (6.05) | 5.95 (4.39)

3. Secondary Outcome: Screen for Child Anxiety Related Emotional Disorders - Parent Version
Description: The Screen for Child Anxiety Related Emotional Disorders - Parent Version (SCARED-P) assesses anxiety symptom severity in youth ages 6-17 years. The parent rates youth anxiety symptoms on 41 items; each item is rated from 0 to 2. Total scores range from 0 to 82, with higher scores indicating greater anxiety severity.
Time Frame: post-treatment (within one week of completing the final of 8 semi-weekly sessions of Attention Bias Modification)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Bias Modification | Placebo Attention Task
Number analyzed (Participants) | 31 | 30
units on a scale | 22.22 (14.23) | 18.05 (12.49)

4. Secondary Outcome: Screen for Child Anxiety Related Emotional Disorders - Child Version
Description: The Screen for Child Anxiety Related Emotional Disorders - Child Version (SCARED-C) assesses anxiety symptom severity in youth ages 6-17 years. The child rates his or her anxiety symptoms on 41 items; each item is rated from 0 to 2. Total scores range from 0 to 82, with higher scores indicating greater anxiety severity.
Time Frame: post-treatment (within one week of completing the final of 8 semi-weekly sessions of Attention Bias Modification)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Bias Modification | Placebo Attention Task
Number analyzed (Participants) | 31 | 30
units on a scale | 14.15 (12.78) | 12.83 (13.60)

5. Secondary Outcome: Screen for Child Anxiety Related Emotional Disorders - Parent Version
Description: as for outcome 3
Time Frame: 8-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Bias Modification | Placebo Attention Task
Number analyzed (Participants) | 24 | 23
units on a scale | 21.05 (14.12) | 17.98 (13.16)

6. Secondary Outcome: Screen for Child Anxiety Related Emotional Disorders - Child Version
Description: as for outcome 4
Time Frame: 8-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Attention Bias Modification | Placebo Attention Task
Number analyzed (Participants) | 24 | 23
units on a scale | 17.75 (16.45) | 12.09 (12.18)

ADVERSE EVENTS:
Time Frame: Duration of study participation (12 weeks on average)
Arm/Group | Attention Bias Modification | Placebo Attention Task
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/31
Other Adverse Events (participants affected / at risk) | 0/33 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Attention Bias Modification (N=33) | Placebo Attention Task (N=31)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) — 9 days after completion of the study protocol, we learned that a participant experienced suicidal ideation and was evaluated at a hospital emergency department. This event was deemed unrelated to the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/11/NCT01819311/Prot_SAP_001.pdf
  • Informed Consent Form (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT01819311/ICF_002.pdf